CLINICAL TRIAL: NCT04174352
Title: A Pilot Study of FES Imaging to Optimize Tamoxifen Dose for Metastatic Breast Cancer Patients With ESR1 Mutations
Brief Title: FES Imaging to Optimize Tamoxifen for Metastatic Breast Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW19046; 2019-0935 (Other: Institutional Review Board); A534260 (Other: UW Madison); SMPH/MEDICINE/MEDICINE (Other: UW Madison); Protocol Ver v.5.0 1/8/2024 (Other: UW Madison); AAH4731 (Other Grant/Funding Number: Multiple donors); NCI-2019-07924 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2019-11-21; First posted 2019-11-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: ERα+ Breast Cancer; ESR1 Gene Mutation
MeSH Terms: interventions — Tamoxifen

STUDY DESIGN:
Intervention Model Description: a single-arm, open-label, pilot study of escalating doses of tamoxifen
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tamoxifen Dose Levels (Experimental): Three participants will be enrolled to each dose level of oral tamoxifen (n = 12)
  Dose Level 1 = 20 mg daily Dose Level 2 = 80 mg daily Dose Level 3 = 160 mg daily Dose Level 4 = 200 mg daily
  Tamoxifen should be started within 14 days of the FES-PET/CT scan, at least 24 hours after FES injection. Participants will continue tamoxifen therapy until there is radiologic or clinical evidence of progressive disease or drug intolerance.
  Interventions: Drug: Tamoxifen; Diagnostic Test: FES PET/CT

INTERVENTIONS:
Drug: Tamoxifen — estrogen modulator
Diagnostic Test: FES PET/CT — Radiolabeled estrogen [18F]-fluoroestradiol (FES) in combination with Positron Emission Tomography / Computed Tomography is a molecular imaging technique for measuring pharmacodynamic effects of endocrine therapy. The injected dose of 18F-FES will be 6 mCi (185 MBq) ± 20% with a specific activity greater than 170 Ci/mmol at the time of injection for an activity dose of 6 mCi. Participant will receive baseline imaging and repeat imaging after 3-4 weeks to evaluate for FES blockade as assigned dose level.

SUMMARY:
Despite broad advancements in endocrine therapy for ERα+ breast cancer, resistance ultimately develops. A common driver of resistance are known ESR1 mutations that lead to constitutively active receptor signaling and transcriptional regulation that is always "turned on" despite the absence of estrogen. Patients with ESR1 mutations are expected to have decreased binding affinity for tamoxifen and thus may be underdosed on standard therapy. [18F]-fluoroestradiol Positron Emission Tomography/Computed tomography (FES-PET/CT) imaging is a novel functional imaging technique that can non-invasively measure ERα expression and inhibition in metastatic ERα+ breast cancer. The proposed a pilot study uses FES-PET/CT imaging to measure ERα blockade to determine the optimal dose of tamoxifen in patients with ESR1 mutations.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed breast cancer that is metastatic or unresectable with the following:

  * Estrogen receptor expression by immunohistochemistry greater than or equal to 10%
  * ESR1 mutation identified using a Clinical Laboratory Improvement Amendments (CLIA) certified assay via tumor biopsy tissue or circulating free DNA (cfDNA)
  * human epidermal growth factor receptor 2 (HER2) negative
* Participants must have measurable disease as defined by RECIST 1.1 or evaluable bone disease with at least one lesion measuring 10 mm or greater in size. (Participants with bone and non-bone disease are eligible. One disease site must meet either the measurable or evaluable criteria outlined.) Participants with liver-only disease are not eligible due to the inherent hepatic uptake related to the radiopharmaceutical's hepatobiliary route of elimination.
* Participants must have received at least 1 prior line of endocrine therapy in the metastatic setting or have had progression within 12 months of adjuvant endocrine therapy. Prior Tamoxifen is allowed in any setting. Prior CDK4/6 in the metastatic setting per NCCN guidelines is allowed.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (See Appendix A)
* Life expectancy of greater than 12 weeks.
* Ability to take oral medications.
* Informed consent: participant must be informed of the investigational nature of the study and must be able to sign a written informed consent.
* Participants with central nervous system (CNS) metastases must be stable after therapy for CNS metastases (such as surgery, radiation, or stereotactic radiosurgery) for at least 1 month.
* Participants must have adequate normal organ and bone marrow function as defined below:

  * Absolute neutrophil count >/= 1,000/mcL
  * Hemoglobin >/= 9.0 g/dL
  * Platelets >/= 100,000/mcL
  * Total bilirubin </= 1.5 x upper limit of normal (ULN)
  * AST (SGOT)/ ALT (SGPT) </= 2.5 x ULN; </= 5 x ULN in the setting of metastatic liver disease
  * Creatinine </= 1.5 x ULN or creatinine clearance >/= 50 mL/min

Exclusion Criteria:

* Prior chemotherapy, radiotherapy, targeted, immunotherapy or investigational therapy within 2 weeks or major surgery within 4 weeks of study enrollment or those who have not recovered (to grade ≤ 1 or baseline) from clinically significant adverse events due to agents administered more than 2 weeks earlier (alopecia and fatigue excluded).
* Participants must not be receiving an ER blocking endocrine therapy (includes fulvestrant, tamoxifen, toremifene, raloxifene) and must be off the agents for a minimum of 60 days prior to planned FES PET/CT to allow for adequate uptake of FES.
* History of allergic reactions attributed to compounds of chemical or biologic composition similar to those of tamoxifen or [18F]-fluoroestradiol.
* Peripheral neuropathy of severity greater than grade 1.
* Current optic nerve disorders, retinopathy, lattice degeneration, macular degeneration, retinal vascular disorder, or retinal tears of severity greater than grade 1.
* History of cerebellar disorders, ataxia, and uncontrolled seizures unless related to transient medical condition and in investigator's opinion is not an active medical issue.
* History of venous thrombosis/thromboembolic event, including pulmonary embolism and stroke.
* Have a heart-rate corrected QT interval (using Fridericia's formula) (QTcF) ≥ 470msec or other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, chronic hypokalemia, family history of long QT interval syndrome).
* Are taking medications that are known to prolong the QT interval, unless they can be transferred to other medications ≥ 5 half-lives prior to dosing or unless the medications can be properly monitored during the study. If equivalent medication is not available, QTcF should be closely monitored.
* Tamoxifen has demonstrated vaginal bleeding, birth defects and fetal loss in pregnant women. Tamoxifen use during pregnancy may have a potential long-term risk to the fetus of a Diethylstilbestrol syndrome (DES)-like syndrome. Women of childbearing potential (WOCP) must not be pregnant (confirmed by a negative urine/serum pregnancy test within 14 days of tamoxifen treatment). In addition, a medically acceptable method of birth control must be used such as an intrauterine device (IUD), use of a double barrier method (condoms, sponge, diaphragm, or vaginal ring with spermicidal jellies or cream), or total abstinence during the study participation and for 3 months after last dose of study drug. Women who are postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) are not considered to be WOCP.
* Ongoing treatment with other investigational agents. Participants cannot be receiving concomitant chemotherapy, radiotherapy, experimental therapy or any other therapy not otherwise outlined by the trial for the purposes of anti-cancer treatment.
* History of uterine malignancy unless participant has had hysterectomy with no evidence recurrent disease for ≥ 3 years from definitive therapy.
* Concurrent malignancy except for the following:

  * Basal cell or squamous cell skin cancer
  * In situ cervical cancer
* The following medications are contraindicated or must be used with caution.

  * Contraindicated:

    * CYP2D6, CYP3A4, and CYP2C9 strong inhibitors
    * CYP2D6, CYP3A4, and CYP2C9 strong inducers
  * Use with caution:

    * CYP2C9 sensitive substrates
    * CYP2D6 moderate inhibitors or inducers
    * CYP3A4 moderate inhibitors or inducers

Note: Transdermal products designed for systemic delivery must be assessed for interaction potential. Topical products not designed to provide systemic delivery (including inhaled products, ophthalmologic products and transvaginal preparations) do not need to be considered.

Contraindicated medications are not allowed. Participants taking these concurrent medications are ineligible unless they can discontinue or switch to alternative medications prior to initiation of study drug (at least 5 half-lives).

Use with caution agents are permitted if a) discontinuation is not feasible or b) no acceptable alternatives are available as determined by the treating physician; however, caution should be used. Consider monitoring by symptoms, labs or drug levels and dose adjustments of the medication.

* Uncontrolled intercurrent clinically significant illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Rate of FES Blockade at each dose level to determine the Optimal Tamoxifen Dose | up to 6 weeks to compare baseline and treatment images
  Reduction in FES uptake will be described and analyzed by Fisher's exact test. Rates or proportion of responses at each dose level will be provided in data listings. If the SUVmax for all 5 target lesions have decreased by > 75% or all 5 lesions have SUVmax<1.5 on the second scan, then these participants will be prospectively defined as having complete FES blockade. If the SUVmax for any of the 5 lesions has not decreased by > 75% or if any new lesions arise with SUVmax ≥1.5, then these subjects will be defined as having incomplete FES blockade.

SECONDARY OUTCOMES:
FES uptake at each dose level: SUVmax | up to 6 weeks to compare baseline and treatment images
  FES uptake will be quantified on 5 target lesions using standardized uptake value (SUV) measurements including SUVmax, SUVmean, SUVpeak, Tumor-to-Normal (T/N) tissue ratio, and Tumor-to-Blood Pool ratios.
FES uptake at each dose level: SUVmean | up to 6 weeks to compare baseline and treatment images
  FES uptake will be quantified on 5 target lesions using standardized uptake value (SUV) measurements including SUVmax, SUVmean, SUVpeak, Tumor-to-Normal (T/N) tissue ratio, and Tumor-to-Blood Pool ratios.
FES uptake at each dose level: Tumor-to-Normal tissue ratio | up to 6 weeks to compare baseline and treatment images
  FES uptake will be quantified on 5 target lesions using standardized uptake value (SUV) measurements including SUVmax, SUVmean, SUVpeak, Tumor-to-Normal (T/N) tissue ratio, and Tumor-to-Blood Pool ratios.
FES uptake at each dose level: Tumor-to-Blood Pool ratio | up to 6 weeks to compare baseline and treatment images
  FES uptake will be quantified on 5 target lesions using standardized uptake value (SUV) measurements including SUVmax, SUVmean, SUVpeak, Tumor-to-Normal (T/N) tissue ratio, and Tumor-to-Blood Pool ratios.
Objective Response Rate at each dose level | up to 6 months
  The objective response rate is the proportion of all participants with confirmed Partial Response or Complete Response according to RECIST 1.1, from the start of treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the start of treatment).
Safety: Number of Participants Experiencing Grade 3 or higher Adverse Events | Up to 21 days on treatment (up to 6 weeks on study)
  All grade 3-4 adverse events occurring between cycle 1, day 1 to cycle 2 day 1 and at least possibly related to therapy will be reviewed by the principal investigator prior to starting enrollment in the next dose cohort. If 2 or more of the 3 participants in any cohort experience grade 3-4 adverse events, then dose escalation will be halted.

CONTACTS AND LOCATIONS:
Overall Officials: Kari Wisinski, MD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Wisconsin Oncology Network (WONIX) sites, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No